CLINICAL TRIAL: NCT03667365
Title: Randomized Study for the Optimal Treatment of Symptomatic Patients With Low Gradient Severe Aortic Valve Stenosis and Preserved Left Ventricular Ejection Fraction
Acronym: ROTAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: new US guidelines
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC17_8843_ROTAS; 2018-A02100-55 (Other: N°ID-RCB)
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Aortic Valve Stenosis
Keywords: severe aortic valve stenosis; low gradient; preserved left ventricular ejection fraction; symptomatic patients
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aortic valve replacement (Experimental)
  Interventions: Procedure: aortic valve replacement
- strict clinical surveillance (Active Comparator)
  Interventions: Other: strict clinical surveillance

INTERVENTIONS:
Procedure: aortic valve replacement — aortic valve replacement surgical or transcatheter aortic valve replacement (will be decided by the heart team before randomization)
  Arms: aortic valve replacement
Other: strict clinical surveillance — strict clinical surveillance strategy
  Arms: strict clinical surveillance

SUMMARY:
According to current European Recommendations on valvular heart disease (VHD), "classical" severe aortic stenosis (AS) is defined by an aortic valve area (AVA) ≤1 cm2 and indexed AVA ≤0.6 cm2/m2, a mean aortic pressure gradient (MAG) >40 mmHg, and a maximal aortic velocity >4 m/sec.

Aortic valve replacement (AVR) is recommended (class I indication) in patients with "classical" severe AS who have any symptoms related to aortic valve disease.

In 2007, Hachicha et al. described a particular pattern of severe AS, characterized by an AVA ≤0.6 cm2/m2, low mean pressure aortic gradient (MAG <40 mmHg), despite the presence of a preserved left ventricular ejection fraction (LVEF ≥50%). This pattern of AS is encountered in nearly 15-25 % of patients who have severe AS. Typically, these patients are elderly subjects, with several comorbidities, a small left ventricular (LV) cavity with pronounced LV concentric remodeling and a restrictive physiology, leading to a decrease in LV stroke volume despite a preserved LVEF. The diagnosis and management of patients with low gradient severe AS and preserved LVEF are often challenging because:

1. the presence of a "true" severe aortic stenosis should be carefully confirmed by a multi-modality imaging approach;
2. the best therapeutic management (AVR versus conservative strategy) of symptomatic patients with low gradient severe AS and preserved LVEF is not clearly established.

In very recently updated European guidelines on the management of VHD, symptomatic patients with low gradient and low flow severe AS and preserved LVEF have only a class IIa-level C indication for AVR. No specific indications are given for the management of symptomatic patients with low gradient and normal flow severe AS. This lack of indications is clearly attributed to a gap in knowledge which requires further investigations to be filled up.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Symptomatic and severe AS defined by an effective AVA ≤1 cm² and indexed AVA ≤0.6 cm2/m2
3. LVEF ≥50%
4. MAG <40 mm Hg (measure confirmed by the multi-window continuous-wave Doppler interrogation and use of Pedoff probe)
5. Confirmation of the presence of severe AS at DSE and MDCT aortic calcium score
6. Feasibility of AVR by surgery or TAVR according to the "heart team"
7. Signature of an informed consent

Exclusion Criteria:

1. Uncontrolled atrial of ventricular arrhythmias
2. Patient having a life expectancy <1 year, independently from their aortic pathology
3. Coronary artery disease necessitating a percutaneous or surgical revascularisation
4. Presence of a concomitant valve disease needing surgical treatment
5. Patient who are included in another research protocol
6. Protected person (adults legally protected (under judicial protection, guardianship or supervision), person deprived of their liberty, pregnant woman, lactating woman and minor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
time from randomization to first occurrence of any of the components of the composite outcome (adjudicated): all-cause mortality or cardiovascular related hospitalization | during 2 years follow-up

SECONDARY OUTCOMES:
rate of all-cause mortality | 2 years
rate of cardiovascular mortality | 2 years
rate of cardiovascular related hospitalization | 2 years
rate of cerebrovascular events | 2 years
walking distance | 6, 12, 18 and 24 months
  6-minute walking test
NT-proBNP plasma levels | 6, 12, 18 and 24 months
quality of life score | 6, 12, 18 and 24 months
  test EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Elena EG Galli, MD, Principal Investigator — CHU Rennes; Erwan ED Donal, PhD, Principal Investigator — CHU Rennes
Locations (18):
- CHU Liège, Liège, Belgium
- France (17):
  - CHU Amiens - Picardie, Amiens
  - CHU Angers, Angers
  - CHU Brest - Hôpital La Cavale Blanche, Brest
  - APHP - CHU Henri Mondor, Créteil
  - CHU Dijon - Hôpital François Mitterrand, Dijon
  - CHU Lille, Lille
  - CH Bretagne Sud, Lorient
  - APHM - Hôpital La Timone, Marseille
  - Clinique du Millénaire, Montpellier
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes
  - CH Saint-Brieuc, Saint-Brieuc
  - Centre Cardiologique du Nord, Saint-Denis
  - CHU Toulouse - Hôpital Rangueil, Toulouse
  - CHU Tours - Hôpital Trousseau, Tours
  - CHU Nancy, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique - Site de Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No